CLINICAL TRIAL: NCT00965354
Title: Mechanisms of Severe Acute Influenza Consortium (MOSAIC)
Acronym: MOSAIC
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Wellcome Trust (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: CRO1367; 09/H0709/52 (Other: English Research Ethics Committee); 09/MRE00/67 (Other: Scottish Research Ethics Committee)
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Influenza
Keywords: severe; acute; influenza; consortium; swine; flu; influenza A; H1N1; hospital; admission
MeSH Terms: conditions — Influenza, Human; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A) Swabs and secretions from the nose and throat B) Blood C) Sputum D) Urine E) Stool
  In addition, if the patients are having further respiratory sample collection as part of their routine care, for example tracheal aspirates, bronchial lavage and other samples then we would like to take an additional amount of these samples for our research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Influenza diagnosis: Patients admitted to hospital with a suspected or confirmed influenza diagnosis on admission

SUMMARY:
The ultimate goal of this collaborative, intensive study is to discover new and effective treatments and to develop better vaccines that can be used in future outbreaks of Influenza A. By integrating the information that we will gather, we will create a unique overview of how influenza causes illness and what might be done to improve patient management.

DETAILED DESCRIPTION:
Influenza A is one of the best studied viruses, but continues to have a very large impact on human and animal health. In addition to causing outbreaks of winter flu, it sometimes mutates to create a new virus that spreads quickly around the world. It is puzzling that the same virus appears to cause minor or absent symptoms in some people while killing others. Much remains to be understood.

The investigators have assembled an unprecedented group of internationally renowned scientists from England and Scotland who will together focus on studying a few hundred people hospitalised during the current swine flu pandemic. Such a large scale project has never before been attempted, but we are now poised to work together and integrate the many recent advances in biomedical science that relate to understanding how influenza causes disease.

ELIGIBILITY:
Inclusion Criteria:

* Any patient admitted to hospital with suspected or confirmed influenza infection

Exclusion Criteria:

* Patients who do not give their consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital admissions
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter JM Openshaw, Principal Investigator — Imperial College London
Locations (8):
- United Kingdom (8):
  - Alder Hey Children's Foundation NHS Trust, Liverpool
  - Royal Liverpool University Hospital, Liverpool
  - Liverpool Women's NHS Foundation Trust, Liverpool
  - Aintree Hospitals NHS Trust, Liverpool
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Royal Brompton and Harefield NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Wirral University Teaching Hospital NHS Foundation Trust, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dunning J, Blankley S, Hoang LT, Cox M, Graham CM, James PL, Bloom CI, Chaussabel D, Banchereau J, Brett SJ, Moffatt MF, O'Garra A, Openshaw PJM; MOSAIC Investigators. Progression of whole-blood transcriptional signatures from interferon-induced to neutrophil-associated patterns in severe influenza. Nat Immunol. 2018 Jun;19(6):625-635. doi: 10.1038/s41590-018-0111-5. Epub 2018 May 18. PMID 29777224
- [Result] Dunning J, Blankley S, Hoang LT, Cox M, Graham CM, James PL, Bloom CI, Chaussabel D, Banchereau J, Brett SJ; MOSAIC Investigators; Moffatt MF, O'Garra A, Openshaw PJM. Author Correction: Progression of whole-blood transcriptional signatures from interferon-induced to neutrophil-associated patterns in severe influenza. Nat Immunol. 2019 Mar;20(3):373. doi: 10.1038/s41590-019-0328-y. PMID 30728492

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Influenza Diagnosis
Started | 131
Completed | 131
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Influenza Diagnosis
Number analyzed (Participants) | 131
Age, Continuous [Mean (Full Range); unit: years] | 42 [17 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 68
Region of Enrollment [Number; unit: participants]
  United Kingdom | 131

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinical Phenotype Presenting Also a Sequential Activation of Immune/Infammatory Pathways.
Description: Detailed clinical phenotype. Clinicopathological correlation will then be sought between the clinical phenotype and pathological parameters measured as per work packages.
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Diagnosis
Number analyzed (Participants) | 131
Participants | 131

ADVERSE EVENTS:
Arm/Group | Influenza Diagnosis
All-Cause Mortality (participants affected / at risk) | 0/131
Serious Adverse Events (participants affected / at risk) | 0/131
Other Adverse Events (participants affected / at risk) | 0/131

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No